CLINICAL TRIAL: NCT02268201
Title: A Randomized, Open-label, Multi-center Clinical Trial to Compare Efficacy and Safety of Cyclosporine-based and Switching Cyclosporine to Tacrolimus of Two Forms-based Immunosuppressive Therapy in Renal Transplant (KTx) Recipients
Brief Title: A Study to Evaluate the Efficacy and Safety in Kidney Transplant Recipients When Changed From Cyclosporine to Tacrolimus Prolonged-release Capsule or Tacrolimus Capsule
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to difficulty enrolling patients
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNKTxCon
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplant Recipients
Keywords: tacrolimus; immunosuppressive therapy
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADV group (Experimental): Once daily
  Interventions: Drug: Advagraf
- PRG group (Experimental): Twice daily
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: Tacrolimus prolonged-release capsule
  Arms: ADV group
Drug: Prograf — oral
  Other Names: Tacrolimus capsule
  Arms: PRG group

SUMMARY:
KTx recipients receiving cyclosporine-based immunosuppressive therapy, and in the opinion of the investigator would benefit from switch to a tacrolimus-based immunosuppression, will switch the immunosuppressive therapy to a tacrolimus-based one. Efficacy and safety of patients will be observed for 52 weeks.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the adherence of kidney transplant recipients treated with Prograf and Advagraf regimens.

The secondary objectives of this study are:

* To compare the renal function (eGFR) in KTx recipients treated with Cyclosporine and Tacrolimus regimens.
* To compare the QoL of KTx recipients treated with Cyclosporine and Tacrolimus regimens.
* To compare the efficacy of Cyclosporine and Tacrolimus regimens in KTx recipients.
* To compare the safety of Cyclosporine and Tacrolimus regimens in KTx recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients have received cyclosporine-based immunosuppressive therapy for more than 6 months， and have maintained a stable regimen for at least 8 weeks before enrollment
* The trough blood level of cyclosporine maintained at 50-200ng/ml at least 4 weeks before enrollment
* SCr< 200 μmol/l ( 2.3 mg/dl)
* Females of childbearing potential must have a negative pregnancy test within 48 hrs prior to randomization and reliable methods of contraception should be started 4 weeks prior to and during the whole study
* Understand and sign the approved informed consent form

Exclusion Criteria:

* Patients who have had other solid organ transplantations
* 24 hours proteinuria>2g
* SGPT/ALT，SGOT/AST or total bilirubin rising to more than double the normal level
* Patients suffering from serious infection lesions
* Patients have severe diarrhea or vomiting, peptic ulcer and/or defective absorption
* Patients have severe heart, lung disease, abnormal glucose tolerance or malignant tumor history
* Known contraindication to administration of Tacrolimus. Subject has known hypersensitivity to tacrolimus, or any of the product excipients
* Pregnancy or lactating women
* Patients have participated in another clinical trial in the past month
* Patient refuses to sign informed consent form
* Patient not willing to continue in the study and wants to withdraw from the study
* Poor adherence or lost to follow-up
* Violation of protocol
* Severe adverse events occurred need to withdraw the study according to investigator's judgment
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
medication adherence | Up to 52 weeks after switching
  VAS will be used to evaluate adherence between PRG and ADV

SECONDARY OUTCOMES:
endogenous creatinine clearance rate (Ccr) | Day 0, Week-1, Week2, Week-4, Week-8, Week-16, Week-24, Week36 and Week-52
Calculated glomerular filtration rate | Day 0, Week-1, Week2, Week-4, Week-8, Week-16, Week-24, Week36 and Week-52
blood lipids | Day 0, Week-1, Week2, Week-4, Week-8, Week-16, Week-24, Week36 and Week-52
  total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol and triglyceride
liver function (AST, ALT and bilirubin) | Day 0, Week-1, Week2, Week-4, Week-8, Week-16, Week-24, Week36 and Week-52
fasting blood-glucose (FBG) | Day 0, Week-1, Week2, Week-4, Week-8, Week-16, Week-24, Week36 and Week-52
Safety assessed by the incidence and severity of adverse events | Up to 52 weeks after switching

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- China (7):
  - Beijing
  - Fuzhou
  - Guangzhou
  - Jinan
  - Nanchang
  - Shanghai
  - Xi'an

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=124